CLINICAL TRIAL: NCT05891587
Title: Semaglutide Therapy for Alcohol Reduction - Tulsa
Acronym: STAR-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: National Institute of Drug Abuse (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202208
Record Dates: First submitted 2023-05-04; First posted 2023-06-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Ozempic; Wegovy; Semaglutide; Addiction; Substance Use; Alcohol drinking; Alcohol-Related Disorders
MeSH Terms: conditions — Alcoholism; Behavior, Addictive; Substance-Related Disorders; Alcohol Drinking; Alcohol-Related Disorders | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Randomized, between-subject, double-blind, and placebo-controlled.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive subcutaneous injections of semaglutide in escalating doses (.25mg to 1.0mg) over the course of 12 weeks.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive subcutaneous injections of a placebo saline solution over the course of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide pen injector
  Arms: Semaglutide
Drug: Placebo — Saline solution
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine if semaglutide, when compared to placebo, is safe and may reduce alcohol drinking in individuals who endorse symptoms consistent with alcohol use disorder.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical trial assessing the efficacy and tolerability of semaglutide in individuals who meet criteria for alcohol use disorder. Participants will complete a remote phone screening and an on-site screening visit to determine study eligibility. Eligible participants will be randomized to receive weekly subcutaneous injections of either semaglutide or a placebo (1:1 ratio). Doses will be titrated according to the FDA-approved dosing schedule starting at a dose of 0.25 mg/week for four weeks, then 0.5 mg/week for four weeks, and finally the dose will be increased to 1.0 mg/week for four weeks, for a total of 12 weeks of treatment. Participants will be asked to complete experimental procedures at the baseline and endpoint visits (Week 1 and Week 12), which include functional magnetic resonance imaging (fMRI) experiments, functional near-infrared spectroscopy (fNIRS) experiments, and virtual reality experiments. Participants will also complete questionnaires, biospecimen collections, and computer-based behavioral therapy modules at various study timepoints. Participants will periodically meet with a study physician and will be monitored for any adverse events. A remote follow-up assessment will take place 9 weeks after the participant's last dosing visit.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent before any trial-related activities
2. Male or female individuals who are at least 18 years old
3. Alcohol Use Disorder (minimum 2 symptoms on a validated diagnostic tool, e.g., DSM-5 Checklist for Alcohol Use Disorder, the Mini-International Neuropsychiatric Interview (MINI) or the Structured Clinical Interview for DSM Disorders (SCID))
4. Self-reported drinking, according to alcohol TimeLine Follow-Back (TLFB), of > 7 drinks per week for females or > 14 drinks per week for males during the 28-day period prior to screening + at least four days with > 3 drinks for females or > 4 drinks for males during the 28-day period prior to screening.
5. Most recent Clinical Institute Withdrawal Assessment for Alcohol - revised (CIWA-Ar) score is ≤ 10
6. Able to speak, read, write, and understand English
7. Normal or corrected-to-normal (e.g., wearing glasses or contacts) vision and normal or corrected-to-normal (e.g., with the use of a hearing aid) hearing
8. Female participants must be postmenopausal for at least one year, surgically sterile, or practicing a highly effective method of birth control before entry and throughout the study and must have a negative urine pregnancy test at each visit. Examples of birth control methods include (but are not limited to) oral contraceptives or contraceptive implants, barrier methods such as diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms, intrauterine devices, a partner with a vasectomy, or abstinence from intercourse.

Exclusion Criteria:

1. BMI < 25 kg/m2 or BMI ≥ 50 kg/m2
2. Evidence of malnutrition as determined by the Nutrition Risk Screening 2002 (NRS-2002)
3. Most recent blood tests: creatinine ≥ 2 mg/dL, eGFR ≤ 60 mL/min/1.73 m2, triglycerides > 500 mg/dl, ALP > 4x the upper normal limit, abnormal blood lipase levels
4. Present diagnosis of diabetes or blood hemoglobin A1c (HbA1c) ≥ 6.5 %
5. Current use of the following medications with glucose lowering properties: GLP-1 analogues, sulfonylurea, insulin, metformin, thiazolidinediones (TZD), dipeptidyl peptidase-4 (DPP-IV) inhibitors, sodium-glucose cotransporter-2 (SGLT-2) inhibitors
6. Current or prior use of semaglutide (Ozempic or Wegovy) or tirzepatide (Mounjaro).
7. Use of weight-lowering/anti-obesity medications within the past 90 days prior to enrollment in the study.
8. Current use of FDA-approved pharmacotherapy for AUD (acamprosate, disulfiram, naltrexone), or other medications that are used for AUD treatment including topiramate and bupropion. Due to the half-life of injectable naltrexone, we will exclude participants who have taken vivitrol in the past 30 days.
9. Current use of medications with known interactions with semaglutide
10. Personal or family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
11. Known history of alcoholic ketoacidosis, pancreatitis (either acute or chronic), pancreatic carcinoma, gallbladder disease, jaundice, Mallory-Weiss syndrome (esophageal tears secondary to vomiting), esophageal varices, cirrhosis
12. Known history of gastric bypass surgery
13. Known or suspected allergy to semaglutide, any of the product components, or any other GLP-1 analogue
14. Known history of suicidal attempts (within the past 24 months) or active suicidal ideation
15. Known history of vestibular disorders or clinically significant motion sickness
16. Known history of noise-induced hearing loss or tinnitus
17. Only for subjects undergoing brain scan: contraindication(s) for brain fMRI
18. Unstable cardiovascular conditions (e.g., arrhythmias, clinically significant ECG abnormalities)
19. Physical and/or mental health conditions that are clinically unstable, as determined by the study clinicians, including (but not limited to) major depressive disorder or generalized anxiety disorder unstable within the past three months or other psychiatric conditions (e.g., schizophrenia, bipolar disorder) unstable within the past twelve months.
20. Current stimulant or opioid use disorder.
21. Any other reason or clinical condition that the Investigators judge would interfere with study participation and/or be unsafe for a possible subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in alcohol drinks per drinking day. | Baseline (Week 1) to post-medication (Week 13)
  The average number of standard alcohol-containing drinks consumed per drinking day (DDD) measured over the 28 days preceding the study baseline visit, and the average DDD during at least the first 14 days at each dose, up to the first 28 days at each dose.

SECONDARY OUTCOMES:
Change in drinks per week. | Baseline (Week 1) to post-medication (Week 13)
  The average number of standard alcohol-containing drinks consumed per week (DPW) measured over the 28 days preceding the study baseline visit, and the average daily consumption during at least the first 14 days at each dose, up to the first 28 days at each dose.
Change in heavy drinking days per week. | Baseline (Week 1) to post-medication (Week 13)
  The average number of heavy drinking days per week measured over the 28 days preceding the study baseline visit, and the average number of heavy drinking days per week during at least the first 14 days at each dose, up to the first 28 days at each dose.
Safety and tolerability of semaglutide in individuals with alcohol use disorder (AUD) | Baseline (Week 1) to post-medication (Week 13)
  Number and grade of adverse events in individuals with AUD who receive semaglutide or placebo
Reduction and/or changes in food choices in a virtual reality buffet-like laboratory | Baseline (Week 1) to post-medication (Week 13)
  Difference in the macronutrient content selected in the virtual reality buffet
Change in blood phosphatidylethanol (PEth) levels as a biomarker of alcohol use | Baseline (Week 1) to post-medication (Week 13)
  Difference in blood PEth levels
Changes in brain activity in response to alcohol cues during fMRI cue reactivity task | Baseline (Week 1) to post-medication (Week 13)
  Group differences in fMRI blood oxygenation level dependent (BOLD) signal within reward neurocircuitry in response to alcohol and nonalcoholic beverage stimuli
Changes in brain activity during an fMRI interoceptive attention task | Baseline (Week 1) to post-medication (Week 13)
  Group differences in fMRI blood oxygenation level dependent (BOLD) signal within interoceptive brain regions during an interoceptive attention task.
Changes in brain activity during an alcohol-related Go/No-Go fNIRS task | Baseline (Week 1) to post-medication (Week 13)
  Difference in activity of inhibitory brain regions during an alcohol-related Go/No-Go fNIRS task.

CONTACTS AND LOCATIONS:
Overall Officials: William K Simmons, Ph.D., Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- OSU Biomedical Imaging Center, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other investigators upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available following publication of study manuscripts and will be available indefinitely.
Access Criteria: Reasonable request from qualified investigator.

REFERENCES:
- See also: Link to online eligibility screener — http://redcap.link/startstudy